CLINICAL TRIAL: NCT06015399
Title: Methods of Establishing Intersegmental Plane in Segmentectomy: a Prospective Randomized Controlled Study
Brief Title: Methods of Establishing Intersegmental Plane in Segmentectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Liu Wenliang, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYF2023098
Record Dates: First submitted 2023-08-20; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Surgery
Keywords: segmentectomy; intersegmental plane; closed insufflation technique; dilatation and collapse technique; randomized controlled study
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed insufflation technique group (Experimental): Closed insufflation technique is characterized by ligation in the proximal portion of targeted bronchus and gas injection in the distal portion. Closed insufflation technique group includes patients undergoing segmentectomy using closed insufflation technique.
  Interventions: Procedure: Implementation of closed insufflation technique during segmentectomy
- Dilatation and collapse technique (Active Comparator): Dilatation and collapse technique is characterized by pure oxygen dilatation and subsequent collapse after the division of targeted bronchus. Dilatation and collapse technique group includes patients undergoing segmentectomy using Dilatation and collapse technique.
  Interventions: Procedure: Implementation of dilatation and collapse technique during segmentectomy

INTERVENTIONS:
Procedure: Implementation of closed insufflation technique during segmentectomy — After the identification the targeted segmental bronchus during the operation,ligating the proximal end of the targeted bronchus. Put the vessel separation forceps in the distal bronchial space to avoid the accidental damage of the vessels. Use a 50ml syringe to inject air into the distal bronchus (about 100ml is expected) until the intersegmental plane is satisfactory. Divide the target bronchus using the cutting and closing device.
  Arms: Closed insufflation technique group
Procedure: Implementation of dilatation and collapse technique during segmentectomy — Divide the target bronchus using the cutting and closing device. Ask the anesthesiologist to inflate the lung completely from pure oxygen to the affected side and then change to single lung ventilation. Wait for the intersegmental plane to appear(usually about 15 minutes).
  Arms: Dilatation and collapse technique

SUMMARY:
The aim of this study is to perform a prospective, single-center, randomized controlled study to explore whether closed insufflation technique is not inferior to dilatation and collapse technique in segmentectomy, and to provide a new option for establishing intersegmental plane in segmentectomy.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized controlled study. A total of 200 subjects undergoing segmentectomy are scheduled to be enrolled within 1 year, and the subjects are randomly divided into closed insufflation group or dilatation and collapse group using a random number table generated by the computer, with 100 cases in each group. Intersegmental plane resolution grading, perioperative complications, operative time, intraoperative blood loss, postoperative hospitay stay, and pulmonary function 3 months and 1 year after surgery will be extracted and compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily join and sign a written informed consent;
2. The age of the subjects is 18-75 years old, regardless of gender;
3. The ECOG PS was 0 or 1;
4. Three-dimensional visualization was performed before surgery, and the surgeon judged that the tumor could be completely removed by segmentectomy, and surgical margin was expected to be greater than 2cm or the maximum diameter of the nodule;
5. Thin-slice CT suggests any of the following: ① The diameter of pulmonary nodules is 2-3cm and the consolidation-tumor ratio (CTR) is less than 0.25; ② Pulmonary nodule diameter ≤2cm and 0.25 < CTR < 0.5; ③ Non-peripheral pulmonary nodule diameter ≤2cm and CTR≤0.25;
6. cN0 and no distant metastasis;
7. Intraoperative freezing examination or postoperative paraffin examination suggest early lung adenocarcinoma;
8. Intraoperative freezing disease of station 12 lymph nodes showed no cancer metastasis;
9. Preoperative anesthesia risk assessment: American Society of Anesthesiologists (ASA) Level I-III;
10. Has no history of lung resection;
11. Has not received anti-tumor therapy such as radiotherapy, chemotherapy, targeted therapy and immunotherapy.

Exclusion Criteria:

1. The subject did not understand the study protocol, did not cooperate or refused to sign the informed consent;
2. The subject has a history of malignant tumor or has previously received anti-tumor therapy;
3. 3D visualization was not received before surgery;
4. The surgeon judged that segmentectomy could not ensure complete resection of the tumor;
5. has a history of lung resection, or chest trauma or surgery on the affected side of chest cavity;
6. Extensive intraoperative dense thoracic adhesion;
7. Conversion to thoracotomy;
8. Intraoperative frozen examination of intrapulmonary lymph nodes indicated cancer metastasis;
9. Pulmonary nodules are located in the right middle lung;
10. Suffered from chronic bronchitis, emphysema, asthma and other chronic lung diseases;
11. Other conditions unsuitable for inclusion in this study deemed by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Intersegmental plane clarity grading | intraoperatively
  Intersegmental plane clarity will be graded as followed: G1: partial collapse of targeted parenchymal tissue, G2: partial dilatation of non-targeted adjacent tissue, G3: dilatation of targeted tissue and unclearness of intersegmental plane, G4: entire dilatation of targeted tissue and clearness of intersegmental plane.
Surgical complications | Up to 3 months
  Surgical complications will be assessed according to the Society of Thoracic Surgeons database criteria.
Operative time required for segmentectomy | From the dissection of segmental structures to finish of segementectomy
  Operative time required for segmentectomy will be measured as the total minutes from initiation to completion of segmentectomy.
Pulmonary function 3 months and 1 year after surgery | Up to 1 year
  Pulmonary function includes ventilation and diffusion function. Pulmonary function will be measured at two time points including 3 months and 1 year after surgery.

SECONDARY OUTCOMES:
Intraoperative blood loss | Intraoperatively
  Intraoperative blood loss will be measured as the total volume of blood loss during the operation.
Postoperative hospital stay | Up to 2 weeks
  Postoperative hospital stay will be measured as the number of days between surgery and discharge.
Days of chest tube placement | Up to 2 weeks
  Days of chest tube placement will be measured as the number of days between surgery and chest tube pull-out.
Safety margin | Up to 1 week
  Minimum distance between nodule and every margin can be measured preoperatively by 3D reconstruction tool and intraoperatively by ruler after the targetd segment has been resected.
Volume of targeted parenchymal tissue | Up to 3 days
  Volume of targeted parenchymal tissue will be calculated by 3D reconstruction tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Surgery, Second Xiangya Hospital of Central South University, China, Changsha, Hunan, China